CLINICAL TRIAL: NCT04491864
Title: DWIBS-MRI: An Adjunct to the Traditional Diagnostic Breast Imaging Evaluation
Acronym: DWIBS
Status: Terminated | Type: Observational
Why Stopped: Further funding was not approved for this study
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 018-781
Record Dates: First submitted 2020-07-27; First posted 2020-07-29 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1.1. Primary Objectives

* To determine if MRI DWIBS can accurately identify suspicious lesions previously categorized on mammography and sonography as potentially malignant.
* We will also validate whether DWIBS-MRI ADC values can be used to accurately differentiate benign from malignant lesions. Additionally, because it is not known whether tumor type or growth rate (Ki67 values) will affect our results, we will include these parameters in our analysis.
* Once we validate the use of DWIBS-MRI ADC values to determine malignancy, can we establish an ADC threshold value to decrease the number of false positive biopsies that are performed while still maintaining a zero false negative rate?
* This study will also assess the correlation between ADC values and the Ki-67 proliferative index of malignant lesions.

ELIGIBILITY:
Inclusion Criteria:

* A patient will be eligible for inclusion in this study if she meets all of the following criteria:

  1. >30 years of age
  2. Genetic Female
  3. Suspected diagnosis of BIRADS 4 or BIRADS 5 masses and/or asymmetries greater than 1 centimeter based on standard 2D/3D mammogram and ultrasound imaging.

Exclusion Criteria:

* A patient is ineligible for inclusion in this study if she meets any of the following criteria:

  1. Prior biopsy of suspicious lesion
  2. Breast implants
  3. Prior history of breast cancer
  4. Patient has a pacemaker
  5. Contraindications to use of MRI imaging (metal implants, etc.)
  6. Woman pregnant or lactating
  7. Calcifications as only findings present for a suspicious lesion

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study population under investigation are for participants who are genetically female.
Study Population: Genetically female patients age 30 and greater with suspicious BIRADS 4 or BIRADS 5 masses and/or asymmetries on standard 2D/3D mammogram and ultrasound imaging
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
MRI DWIBS Accuracy | 1 month
  • To determine if MRI DWIBS can accurately identify suspicious lesions previously categorized on mammography and sonography as potentially malignant.
Validate DWIBS-MRI | 1 month
  • We will also validate whether DWIBS-MRI ADC values can be used to accurately differentiate benign from malignant lesions. Additionally, because it is not known whether tumor type or growth rate (Ki67 values) will affect our results, we will include these parameters in our analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White Research Insitute, Dallas, Texas, United States